CLINICAL TRIAL: NCT04711343
Title: A Randomized, Double-blinded, Single-dose, 3-arms Parallel, Comparative Study to Evaluate the Pharmacokinetics and Safety of BAT2306 Injection vs Secukinumab Injection (Cosentyx®) in Healthy Chinese Male Subjects
Brief Title: Comparative Study to Evaluate the Pharmacokinetics of BAT2306 vs Cosentyx® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-2306-001-CR
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAT2306 injection (Experimental): 150mg /1ml; subcutaneous injection
  Interventions: Drug: BAT2306
- Cosentyx (US-licensed) (Active Comparator): 150mg /1ml; subcutaneous injection
  Interventions: Drug: Cosentyx (US-licensed)
- Cosentyx (EU-licensed) (Active Comparator): 150mg /1ml; subcutaneous injection
  Interventions: Drug: Cosentyx (EU-licensed)

INTERVENTIONS:
Drug: BAT2306 — 150mg/1 ml; single dose；prefilled syringe; subcutaneous injection
  Arms: BAT2306 injection
Drug: Cosentyx (US-licensed) — 150mg/1 ml; single dose；prefilled syringe; subcutaneous injection
  Other Names: Secukinumab
  Arms: Cosentyx (US-licensed)
Drug: Cosentyx (EU-licensed) — 150mg/1 ml; single dose；prefilled syringe; subcutaneous injection
  Other Names: Secukinumab
  Arms: Cosentyx (EU-licensed)

SUMMARY:
It is a randomized, double-blinded, single-dose, 3-arm parallel, comparative study to evaluate the pharmacokinetics, safety and immunogenicity of BAT2306 Injection vs Cosentyx® (EU-licensed and US-licensed) in healthy Chinese male subjects. A total of 216 healthy male subjects are planned to be included and randomized at a ratio of 1:1:1 to receive single 150mg BAT2306 Injection or Cosentyx® (EU-licensed and US-licensed).

DETAILED DESCRIPTION:
The study has a screening period of 14 days. PK blood samples will be collected from subjects to determine the serum concentration of Secukinumab, thus to evaluate the similarity of the pharmacokinetics of the three study drugs.

The investigator will perform safety evaluation for vital signs, physical examinations, injection site reaction, ECG, clinical laboratory tests and adverse events throughout the study. Immunogenicity evaluation (ADA, ADA titration and NAb) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male healthy subjects aged from 18 to 55 years (including the boundary value)；
* BMI between 18-28kg/m2 (including boundary value) and body weight between 55-85kg;
* Normal physical examination results or abnormal with no clinical significance according to the doctor's judgment;
* The subject (including partner) has no pregnancy plan or sperm donation plan during the whole trial period and within 6 months after the completion of the study, and voluntarily adopts effective contraceptive measures;
* Sign the informed consent before joining the study, and fully understand the content, process and possible risks;
* Willing and able to comply with the visits and treatments of the trial protocol.

Exclusion Criteria:

* Clinical laboratory examination results are abnormal and with clinical significance, or other clinical findings indicate diseases (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, tumor, pulmonary, immune, mental or cardiovascular and cerebrovascular diseases) with clinical significance within one year prior to screening；
* ECG is abnormal and has clinical significance (judged by the investigator);
* With active infection within two months before screening, including acute and chronic infection and local infection;
* Hepatitis B and/or Hepatitis C; or HIV antigen/antibody positive; or Treponema pallidum antibody positive;
* Having taken any prescription drug, over-the-counter drug, any vitamin product or herbal medicine within 28 days before screening (or within 5 half-lives of the above drugs, whichever is longer);
* Having participated in drug clinical trials within 3 months before the study administration, or planning to participate in other drug clinical trials during the study period;
* Acute disease occurred or with concomitant medication from the screening to use of the study drug; major injury or surgery or fracture occurred within 4 weeks before enrollment, or surgery was planned during the study;
* Having used Secukinumab (or its biosimilars) or interleukin (IL-17) targeting agents, or having used any biological products or monoclonal antibodies within 3 months before screening (or within 5 half-lives of the drugs, whichever is longer);
* Having received within 12 weeks prior to initiating treatment or planning to receive live vaccines during the study;
* Suspected or confirmed as allergic constitution (allergic to variety of drugs or food), or allergic to Secukinumab, or severe allergic or allergic reaction to monoclonal antibody;
* Blood donation or massive blood loss (> 450 ml) within 3 months before using the study drug, or planning to donate blood during the study, or having received blood transfusion within 8 weeks before screening;
* Positive urine drug screening or drug abuse history or drug use in the past five years;
* Employees or relatives of all investigators, clinical centers, clinical research organizations or sponsors cannot be included in the group;
* Subjects considered unsuitable by the investigators.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Endpoint：Peak plasma concentration (Cmax) | 0-5months
  Pharmacokinetics Endpoint：Peak plasma concentration (Cmax)
Pharmacokinetics Endpoint：Area under the plasma concentration versus time curve (AUC0-inf) | 0-5months
  Pharmacokinetics Endpoint：Area under the plasma concentration versus time

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Principal Investigator — The First Hospital of Jinlin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
Only one site study